CLINICAL TRIAL: NCT01168960
Title: Identifying Multiple Mechanisms of Change in Alcoholism Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Paul Stasiewicz, Senior Research Scientist, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5RC1AA018986 (NIH)
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Cognitive Behavioral Therapy; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cognitive Behavioral Treatment (Other): A single intervention study
  Interventions: Behavioral: Cognitive behavioral therapy for alcohol dependence

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for alcohol dependence — 12-session behavioral treatment that incorporates behavioral skills training targeting high-risk drinking behavior.

SUMMARY:
Cognitive-behavioral therapy (CBT) is an effective treatment for alcohol dependence, but little is known about how CBT works to achieve these effects. Although several possible mechanisms have been proposed to explain the effects of CBT, it is rare that more than one mechanism is studied. However, it may be the case that similar outcomes (e.g., abstinence) may be reached through multiple paths. Therefore, essential to conducting work on behavioral change mechanisms is distinguishing different courses or paths and moderating influences (Kazdin, 2007). In the present study, we will focus on 2 key mechanisms posited to underlie the effectiveness of CBT specifically, increasing self-efficacy and self-confidence and reducing positive outcome expectancies for alcohol use, and 2 key mechanisms posited to underlie the effectiveness of a wide range of therapeutic interventions, increasing the therapeutic alliance and reducing/regulating negative emotional states. For the present study, participants will be 72 alcohol dependent men and women who agree to participate in a 12-week trial of CBT for alcohol dependence. In addition, comprehensive research assessments will be conducted with patients at baseline, end of treatment, and 3-months posttreatment.

Specific Aim 1. To examine the within-treatment week-to-week relationship between ratings of 4 key therapeutic mechanisms and alcohol involvement (operationalized as percent days abstinent {PDA} and drinks per drinking day {DDD}) during treatment. It is hypothesized that self-efficacy, outcome expectancies, therapeutic alliance (as rated by the patient and therapist), and negative affect assessed after any given treatment session will each predict alcohol involvement during the following week. Exploratory analyses also will investigate the relationship of a given week's alcohol involvement on each of the four key variables as assessed the following week.

Specific Aim 2. To examine profiles of the four key mechanisms over the course of treatment in relation to alcohol involvement during treatment and during the 3-month follow-up period. These analyses will be descriptive/exploratory. It is expected that profiles will emerge with the key mechanisms that are associated with decreased alcohol involvement (for example, when the alliance is relatively strong throughout treatment or when the alliance grows stronger over the course of treatment, or when positive outcome expectancies grow weaker over the course of treatment, etc.). Similarly, it is hypothesized that profiles will emerge that are associated with little improvement in alcohol involvement (for example, when negative affect is relatively high throughout treatment or when self-efficacy weakens over the course of treatment).

ELIGIBILITY:
Inclusion Criteria:

* Alcohol Dependent; live within commuting distance of program site; willing to sign informed consent.

Exclusion Criteria:

* Diagnosis of schizophrenia or other psychotic disorder; present with gross neurocognitive impairment; have a current drug use diagnosis other than nicotine or marijuana abuse; have been in substance abuse treatment over the previous 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-01; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Timeline Followback for alcohol | 3-months posttreatment
  Follow-up assessments of drinks per drinking day and percent heavy drinking days will occur at posttreatment and 3-months posttreatment. The timeline followback is a retrospective calendar measure on an individuals self-report of daily alcohol consumption

CONTACTS AND LOCATIONS:
Overall Officials: Paul R. Stasiewicz, Ph.D., Principal Investigator — University at Buffalo
Locations (1):
- Research Institue on Addictions, Buffalo, New York, United States

REFERENCES:
- [Background] Kazdin AE. Mediators and mechanisms of change in psychotherapy research. Annu Rev Clin Psychol. 2007;3:1-27. doi: 10.1146/annurev.clinpsy.3.022806.091432. PMID 17716046